CLINICAL TRIAL: NCT06595550
Title: The Effect of Whey Protein Consumption on Hypoglycemia in Adults with Type 1 Diabetes During the Fasting Holy Month of Ramadan: a Randomized, Crossover Study
Brief Title: The Effect of Whey Protein Consumption on Hypoglycemia in Adults with Type 1 Diabetes During Fasting Ramadan.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ICT23J/001/01
Record Dates: First submitted 2024-01-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Type1 Diabetes; Fasting; Nutrition, Healthy
MeSH Terms: conditions — Fasting | interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- whey protein (Experimental): whey protein with suhoor
  Interventions: Dietary Supplement: Whey protein
- no whey protein (Placebo Comparator): no whey protein with suhoor
  Interventions: Dietary Supplement: no Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Powder milk
  Arms: whey protein
Dietary Supplement: no Whey protein — Powder milk
  Arms: no whey protein

SUMMARY:
Cross over randomized design for adding whey protein to Suhoor meal for patients with T1DM during fasting Ramadan

DETAILED DESCRIPTION:
Patients with type1 diabetes who intend to fast will be supplied with dietary supplement "Whey protein" to be taken with Suhoor (predawn meal) for one week during Ramadan. They will be then crossed over to not taking the whey protein for another week. the order of taking whey protein will be randomized.

During both weeks patients will be monitored through flash continuous glucose monitoring and data will be compared in regards to incidence and timing of hypoglycemia, hyperglycemia, and time in target range.

After Ramadan data will be collected on number of days they had to brake fast due to low blood sugar during both weeks and overall satisfaction with using whey protein during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes Mellitus
2. Age >14 years
3. Committed to do Regular SMBG or on CGM
4. On Multiple Daily Injections or insulin pumps
5. On carbohydrate counting for meal dosing
6. Have previously fasted Ramadan
7. willing to fast Ramadan this year
8. Well-educated about requirements for fasting Ramadan

Exclusion Criteria:

1. Hypoglycemia unawareness
2. Cognitive impairment or learning disability
3. Renal and hepatic impairment
4. Adrenal insufficiency
5. Pregnancy
6. Alcohol consumption
7. Any diagnosed psychiatric disease
8. Sensor-augmented insulin pumps
9. HbA1c >12%
10. Already on protein supplements

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia incidence rate | 1 month
  number of hypoglycemic events (blood glucose <70mg/dl) as detected by flash glucose monitoring

SECONDARY OUTCOMES:
Percentage Time-below-range (TBR), time-above-range (TAR), and time-in-range (TIR) prior to and following whey protein consumption 2. | 1 month
  Glucose profiles as detected by flash glucose monitoring
Glycemic control (HbA1c) and GMI during protein consumption | 1 month
  glucose parameters detected by flash glucose monitoring by and lab
number of days they needed to brake the fast during each week | 1 month
  number of days fast broken during each week
Patient preferences through questionnaire | 1 month
  to compare patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Reem Alamoudi, MD, Principal Investigator — Ministry of National Guard Health Affairs
Locations (1):
- King Abdullah International Research Centre, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No